CLINICAL TRIAL: NCT05806541
Title: The Effect Of Laughter Therapy On Self-Efficacy And Psychological Well-Being İn Nursing Students
Brief Title: The Effect Of Laughter Therapy On Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: sinopUyasemin-1
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Laughter; Self Efficacy
Keywords: laughter therapy; self efficacy; nursing student; well being
MeSH Terms: conditions — Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): At the beginning of the study, data collection tools Personal Information Form, Academic Self-Efficacy Scale and Psychological Well-Being Scale will be applied to the control group. No intervention will be made in the control group. Measurement tools will be applied for the post-test.
- experimental group (Experimental): Arm: Experimental: experimental group Personal Information Form, Academic Self-Efficacy Scale and Psychological Well-Being Scale will be applied to all 4th year nursing students studying at Sinop University Health Sciences in the autumn term of 2023-2024.
  Laughter therapy session will be applied face to face for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. Psychological Well-Being Scale and Academic Self-Efficacy Scale will be applied again after the application and in the follow-up (after the application is over).
  Interventions: Behavioral: laughter therapy

INTERVENTIONS:
Behavioral: laughter therapy — Laughter therapy session will be applied online for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. In the laughter therapy session, the practices of introducing the practitioner and introducing the therapy, breathing exercises for a healthy life, keeping the rhythm accompanied by music, turning the laughter that started as if it were childlike games into reality will be carried out.
  Arms: experimental group

SUMMARY:
Brief Summary: Laughter is an innate, universal response we give to events in our lives. "Laughter Therapy" is a technique created by combining breathing techniques and laughter and takes its place in complementary medicine. It is a simulation performed by making eye contact with the members of the group, in which physical exercise and childlike games take place. Laughter sessions are about 30-40 minutes. continues and this simulation in a short time creates a real and contagious laugh. It has been determined by studies that laughter therapy physiologically increases breathing and relaxes muscles, strengthens mental function by decreasing the level of stress hormones, reduces burnout, depression and anxiety levels, positively affects quality of life, increases social interaction and provides psychological well-being.

Self-efficacy, on the other hand, is a state that expresses a person's belief that he or she is able to perform a certain task. More broadly, self-efficacy examines an individual's ability to perform a task rather than individual characteristics such as physical or psychological characteristics. Psychological well-being is as important as self-efficacy in the development of students. In addition, studies on mental health have generally focused on anxiety and depression. Most of these studies were related to well-being and contributed to the literature. Psychological well-being is defined as managing existential challenges in life.

Aim: This study was planned to determine the Effect of Laughter Therapy on Self-Efficacy and Psychological Well-Being in Nursing Students.

DETAILED DESCRIPTION:
Method: This study will be carried out with 3rd and 4th year students studying at Sinop University, Faculty of Health Sciences, Department of Nursing. It is aimed to include all first-year nursing students in the study. The study will be carried out in the autumn semester of the 2023-2024 academic year. The sample of the study will be all young women studying at the Faculty of Health Sciences, meeting the inclusion criteria and agreeing to participate in the study.

Arm Title: Control Group At the beginning of the study, data collection tools Personal Information Form, Academic Self-Efficacy Scale and Psychological Well-Being Scale will be applied to the control group. No intervention will be made in the control group. Measurement tools will be applied for the post-test.

Arm Title: Experimental Group Personal Information Form, Academic Self-Efficacy Scale and Psychological Well-Being Scale will be applied to all 4th year nursing students studying at Sinop University Health Sciences in the autumn term of 2023-2024.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Study as a nursing student at the Faculty of Health Sciences where the study will be conducted,
* Being a nursing first class student,
* Volunteering to participate in the study.
* Absence of any psychological disorder

Exclusion Criteria:

* Not to study as a nursing student at the Faculty of Health Sciences where the study will be conducted,
* Not to comply with the criteria for inclusion in the study and
* Not to volunteer to participate in the study.
* Have any psychological problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | one day
  This form consists of questions such as age, gender, distraction, loss of interest in lessons, eating problems, sleep status, stress, anxiety, fear, social media use.

SECONDARY OUTCOMES:
Academic Self-Efficacy Scale | one day
  The Academic Self-Efficacy Scale (ASES) was developed by Bulfone et al. in 2019 as 14 items and four sub-dimensions to determine the academic self-efficacy of undergraduate nursing students. Sub-dimensions of the scale 1- Intrinsic Emotion Management (items 1, 2, 3) from 3 items, 2-Automatically Controlled Behavior (items 4, 5, 6, 7) consisting of 4 items, 3-External Emotion Management (8, 9, 10) 4-Socialism (items 11, 12, 13) consists of 5 items. The items of this scale are scored with a 5-point Likert type (1=I don't trust myself at all, 5=I have a lot of confidence in myself) in response to the question "How much do you trust yourself". The score of each question varies between 1-5 and consists of positive items. The Cronbach Alpha value of the scale was obtained as 0.84.

OTHER OUTCOMES:
Psychological Well-Being Scale | one day
  It was developed by Diener et al., (2010) and adapted into Turkish by Telef (2013). It is a single factor, 7-point Likert scale consisting of 8 items. The range of scores obtained varies between 8 and 56. The Cronbach alpha internal consistency coefficient obtained in the reliability study of the scale was calculated as .80. The items of the Psychological Well-Being Scale are answered between 1 and 7, as I strongly disagree (1) to I strongly agree (7). All items are expressed positively. Scores range from 8 (strongly disagree to all items) to 56 (strongly agree to all items). A high score indicates that the person has many psychological resources and strengths.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Özyer, PhD, Principal Investigator — Sinop University
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No